CLINICAL TRIAL: NCT00984256
Title: Pilot Evaluation of Weekly Dosing of Atovaquone/Proguanil (Malarone ®) for Malaria Chemoprophylaxis
Brief Title: Weekly Dosing of Malarone ® for Prevention of Malaria
Acronym: MALWEEK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WRAIR 1583; HSRRB # A-15648 (Other: USAMRMC)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Malaria
Keywords: Malaria; Prophylaxis; Atovaquone; Malarone; Challenge
MeSH Terms: conditions — Malaria | interventions — atovaquone, proguanil drug combination; Atovaquone; Human Challenge Trials as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): 5 groups, each group receiving Malarone tablet(s) (250/100mg)prior to challenge.
  Group 1 - 1 tablet 1 day before challenge Group 2 - 1 tablet 4 days before challenge Group 3 - 1 tablet 7 days before challenge Group 4 - 2 tablets 7 days before challenge Group 5 - 4 tablets 7 days before challenge
  Interventions: Drug: Atovaquone Proguanil; Other: Procedure - malaria challenge
- Control -no prophylaxis (Placebo Comparator)
  Interventions: Other: Procedure - malaria challenge

INTERVENTIONS:
Drug: Atovaquone Proguanil — Volunteers will receive doses of atovaquone/proguanil (Malarone) or matching sugar pills.
  Other Names: Malaria; Prophylaxis; Atovaquone; Malarone; Challenge
  Arms: Drug
Other: Procedure - malaria challenge — 2) Procedure- Malaria Challenge- Volunteers will be exposed to bites of infectious mosquitoes with the intention of causing malaria infection. Volunteers infected with malaria will undergo approved treatments for malaria.
  Other Names: Malaria; Prophylaxis; Atovaquone; Malarone; Challenge

SUMMARY:
The purpose of this study is to determine whether Malarone ®, which is a drug approved to prevent malaria when taken daily, will still effectively prevent malaria if taken weekly.

DETAILED DESCRIPTION:
In this study, two groups of volunteers will be exposed to malaria through the bites of infected mosquitoes. In one group, volunteers will be randomly assigned to one of 5 arms. Each of these arms will receive a different dose of Malarone®, a drug known to prevent malaria when taken daily. Each of these doses will be lower than the maximum approved dose of this medicine. The other group will not be treated with any drug that could prevent symptoms or infection.

After exposure, both groups will be monitored for a period of approximately 3 months to see if they develop symptoms of malaria. Any subjects who do so will be treated with appropriate medications. Subjects in both groups will have their blood checked regularly during this period for the presence of malaria parasites. At the completion of the study, results will be analyzed to determine whether any of the doses of Malarone might effectively prevent malaria if taken weekly rather than daily.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant, non-lactating female 18 to 50 years of age (inclusive) at the time of screening
* Free of clinically significant health problems
* Baseline ECG before entering into the study
* Available to participate for duration of study (approximately 4 months, not including screening period)
* If the participant is female, not pregnant or lactating and willing to use contraception to prevent pregnancy
* BMI between 19 and 30

Exclusion Criteria:

* History of malaria or travel to a malarious country within the previous 12 months
* History of participation in a study in which potential exposure to malaria or vaccination against malaria occurred.
* Planned travel to malarious areas during the study period.
* History of malaria chemoprophylaxis within 60 days prior to time of study entry.
* Chronic use of antibiotics with anti-malarial effects
* Chronic use (defined as more than 14 days)of immunosuppressants or other immune-modifying drugs within six months of study entry.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination, ECG or laboratory screening tests
* Significant unexplained anemia
* History of sickle cell disease or sickle cell trait
* Seropositive for hepatitis B or hepatitis C
* History of splenectomy
* Pregnant or lactating female, or female who intends to become pregnant during the study
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV
* History of a neuropsychiatric disorder (anxiety, depression, psychosis, schizophrenia)
* Chronic or active illicit and/or intravenous drug use
* History of allergy to atovaquone, proguanil or chloroquine
* History of psoriasis
* Concurrent participation in other research studies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Deye, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Result] Deye GA, Miller RS, Miller L, Salas CJ, Tosh D, Macareo L, Smith BL, Fracisco S, Clemens EG, Murphy J, Sousa JC, Dumler JS, Magill AJ. Prolonged protection provided by a single dose of atovaquone-proguanil for the chemoprophylaxis of Plasmodium falciparum malaria in a human challenge model. Clin Infect Dis. 2012 Jan 15;54(2):232-9. doi: 10.1093/cid/cir770. Epub 2011 Nov 3. PMID 22052893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were healthy male and non-pregnant or lactating females between the ages of 18 and 50 with a body mass index (BMI)between 19 and 30 for subject receiving the drug.
Groups:
- Control: The six volunteers in control cohort were enrolled as infectivity controls and did not undergo randomization or receive any study drug.
- Malarone Treatment: Within the Malarone Arm, thirty volunteers were randomized into the below 5 treatment groups, each group receiving Malarone tablet(s) (250/100mg)prior to challenge.
  Group 1 - 1 tablet 1 day before challenge Group 2 - 1 tablet 4 days before challenge Group 3 - 1 tablet 7 days before challenge Group 4 - 2 tablets 7 days before challenge Group 5 - 4 tablets 7 days before challenge
Period: Overall Study
Arm/Group | Control | Malarone Treatment
Started | 6 | 30
Completed | 6 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: one subject withdrew consent
Groups:
- Malarone: Thirty (30) subjects were placed in the Malarone (treatment) Arm. The thirty subjects were then randomized into 5 treatment groups, each group receiving Malarone tablet(s) (250/100mg)prior to challenge. The groups received treatment as follows:
  Group 1 - 1 tablet 1 day before challenge Group 2 - 1 tablet 4 days before challenge Group 3 - 1 tablet 7 days before challenge Group 4 - 2 tablets 7 days before challenge Group 5 - 4 tablets 7 days before challenge
- Control: The six (6) Control volunteers were enrolled in a open label arm and received no treatment prior to malaria challenge.
- Total: Total of all reporting groups
Arm/Group | Malarone | Control | Total
Number analyzed (Participants) | 29 | 6 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 6 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 12
  Male | 18 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 29 | 6 | 35

OUTCOME MEASURES:

1. Primary Outcome: Prophylactic Efficacy of 3 Different Doses of Atovaquone/Proguanil (Malarone@) Given 1 Week Before Infectious Sporozoite Challenge Using the P. Falciparum Human Challenge Model.
Description: Number of participants with prophylactic efficacy was determined by the absence of cases of malaria parasitemia, defined as microscopically detectable parasitemia by Giemsa-stained thick smears, in those receiving any dose of Malarone as compared to the control (no treatment) group
Time Frame: Days 6-20
Population: Analysis population was "According to Protocol" which included participants meeting all eligibility criteria, not meeting any elimination criteria, complying with defined protocol procedures and for whom data are available.
Measure: Number; unit: participants with negative parasitemia
Groups:
- Treatment Group 1: (Group 1) Malarone 1 tablet (250/100 mg) orally administered once 1 day prior to challenge
- Treatment Group 2: (Group 2) Malarone 1 tablet (250/100 mg) orally administered once on day 4 after challenge
- Treatment Group 3: (Group 3) Malarone 1 tablets (250/100 mg) orally administered once 7 days prior to challenge
- Treatment Group 4: (Group 4) Malarone 2 tablets (500/200 mg) orally administered once 7 days prior to challenge
- Treatment Group 5: (Group 5) Malarone 4 tablets (1000/400 mg) orally administered once 7 days prior to challenge
- Control: Six volunteers for the control cohort were enrolled as an infectivity control and did not undergo drug dosing.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Control
Number analyzed (Participants) | 6 | 4 | 5 | 6 | 6 | 6
participants with negative parasitemia | 6 | 4 | 3 | 6 | 5 | 0

2. Secondary Outcome: Measured Concentrations of Plasma Atovaquone With Determinations of T1/2.
Description: Plasma concentrations (ng/ml) were used to determine the elimination half life (t1/2) of atovaquone (days).
Time Frame: 7, 6, 5, and 1 day prior to challenge; on the day of the challenge; 1, 4, 5, 6, 7, 8, 10and 14 days after the challenge; and on the day parasitemia develops.,
Population: Population for analysis included According to Protocol Population.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Prophylaxis Group 1: (Group 1) Malarone 1 tablet (250/100 mg) orally administered once 1 day prior to challenge
- Prophylaxis Group 2: (Group 2) Malarone 1 tablet (250/100 mg) orally administered once on day 4 after challenge
- Prophylaxis Group 3: (Group 3)Malarone 1 tablets (250/100 mg) orally administered once 7 days prior to challenge
- Prophylaxis Group 4: (Group 4) Malarone 2 tablets (500/200 mg) orally administered once 7 days prior to challenge
- Prophylaxis Group 5: (Group 5) Malarone 4 tablets (1000/400 mg) orally administered once 7 days prior to challenge
Arm/Group | Prophylaxis Group 1 | Prophylaxis Group 2 | Prophylaxis Group 3 | Prophylaxis Group 4 | Prophylaxis Group 5
Number analyzed (Participants) | 6 | 4 | 5 | 6 | 6
Days | 3.3 (1.9) | 3.3 (1.2) | 3.3 (1.6) | 5.6 (3.1) | 3.7 (1.4)

3. Secondary Outcome: Measured Concentrations of Plasma Atovaquone With Determinations of Area Under the Curve
Description: Plasma concentrations were used to determine the pharmacokinetic curves with determinations of area under the curve (AUC).The smallest AUC Day 0-6.5 associated with protection from detectable parasitemia, and the highest AUC Day 0-6.5 observed in any cases of malaria (prophylactic failures) were to be reported.
Time Frame: as for outcome 2
Population: Analysis was done on subjects who completed the study according to protocol
Measure: Mean (Standard Deviation); unit: ng*day/ml
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5
Number analyzed (Participants) | 6 | 4 | 5 | 6 | 6
ng*day/ml | 3595 (2213) | 616 (191) | 510 (218) | 1434 (664) | 2233 (1895)

ADVERSE EVENTS:
Time Frame: 7 days before challenge until end of the study (Day 90)
Groups:
- Drug: Partially randomized, double-blind, placebo-controlled trial using a human Plasmodium falciparum challenge to evaluate malaria chemoprophylaxis of Malarone in 36 healthy adults. Subjects were enrolled in 1 of 2 cohorts based on subject preference. Thirty subjects were placed in the prophylaxis cohort (Cohort 1) and 6 subjects were placed in the control cohort (Cohort 2)
  5 treatment groups, each group receiving Malarone tablet(s) (250/100mg)prior to challenge.
  Group 1 - 1 tablet 1 day before challenge Group 2 - 1 tablet 4 days before challenge Group 3 - 1 tablet 7 days before challenge Group 4 - 2 tablets 7 days before challenge Group 5 - 4 tablets 7 days before challenge
- Control: no malarone prophylaxis received
Arm/Group | Drug | Control
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/6
Other Adverse Events (participants affected / at risk) | 16/29 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=29) | Control (N=6)
(General disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=29) | Control (N=6)
Headache (Nervous system disorders) | 15 (22) | 2 (2) — Headache was the most common event
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes